CLINICAL TRIAL: NCT03742674
Title: Independence Stairs Climbing Ability Prediction During the Sub-acute Rehabilitation Phase of People After Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: SHEBA-18-5299-OK-CTIL
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: CVA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort patients post stroke
  Interventions: Other: Follow up

INTERVENTIONS:
Other: Follow up — No intervention

SUMMARY:
Independence stairs climbing ability prediction during the sub-acute rehabilitation phase of people after stroke

ELIGIBILITY:
Inclusion Criteria:

* First cerebro vascular accident (CVA) diagnosis
* Basic cognitive and communicative abilities

Exclusion Criteria:

* Traumatic brain injury (TBI)
* Confusion state and lack of cooperation due to brain lesion
* Unstable cardiovascular status
* Independently climbing stairs ability at entrance

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post stroke Age 18-69 years Hospitalized in brain injury rehabilitation at Sheba Tel-Hashomer medical center
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Independently climbing stairs ability | Through study completion, an average of 1-2 years
  Yes / No

SECONDARY OUTCOMES:
Time post stroke | Through study completion, an average of 1-2 years
  Days
Time for ascending and descending staircase | Through study completion, an average of 1-2 years
  Seconds
Stairs climbing tipe | Through study completion, an average of 1-2 years
  Step over / Step to, use of handrail